CLINICAL TRIAL: NCT04411420
Title: Improving Veteran Access to Integrated Management of Back Pain: A Pragmatic, Cluster Randomized Trial
Brief Title: Improving Veteran Access to Integrated Management of Back Pain
Acronym: AIM-BACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Durham VA Medical Center (U.S. Federal Agency); University of North Carolina, Chapel Hill (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00101938; UH3AT009790 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain; Veterans Family
Keywords: clinical pathway; veterans; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This study is a 4-year cluster randomized pragmatic trial comparing the effectiveness of a sequenced, multi-modal integrated care pathway for lower back pain (LBP) to a care management by pain navigator program for LBP. The study target population is veterans seeking services for lower back pain in participating VA clinics.
  We plan to enroll 16 VA clinics randomized in a 1:1 Ratio using a covariate constrained randomization.
Who Masked: Outcomes Assessor
Masking Description: The only blinded members of the project include the VA research and Duke Clinical Research Institute (DCRI) research staff members administering the consent and follow up survey data collection processes. All other team members will be unblinded due to the pragmatic design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Care Pathway (Active Comparator): The integrated care pathway provides both on-site physical therapy services and centrally-delivered services via telephone or video from study providers at the Durham VA.
  Interventions: Behavioral: Pain modulation with physical pain treatment; Behavioral: Telephone delivered self-management counseling for increasing physical activity; Behavioral: Telephone delivered behavioral treatment for participants with high risk for continued disability
- Coordinated Care Management Pathway (Active Comparator): The care management pathway involves a referral of patients from a physician to a pain navigator on site at the local VA who is knowledgeable in current recommended treatment guidelines for low back pain.
  Interventions: Behavioral: Patient preference treatment protocol; Behavioral: Nonpharmacological guideline adherent treatment protocol; Behavioral: Facilitated referrals to existing VA or non-VA pain management resources

INTERVENTIONS:
Behavioral: Pain modulation with physical pain treatment — Examples of pain modulation with physical pain treatment include spinal manipulation, massage, or transcutaneous electrical nerve stimulation
  Arms: Integrated Care Pathway
Behavioral: Telephone delivered self-management counseling for increasing physical activity — Centrally located physical therapy assistants will provide six weeks of telehealth consults to increase physical activity for the patient
  Arms: Integrated Care Pathway
Behavioral: Telephone delivered behavioral treatment for participants with high risk for continued disability — Patients with a higher risk of developing chronic or persistent back pain will be identified using the nine question risk stratification start back screening tool (SBST) and will receive six additional weeks of physical activity instructions and additional pain modulation treatments as needed.
  Arms: Integrated Care Pathway
Behavioral: Patient preference treatment protocol — the pain navigator will work through a shared decision making process with the patient to determine the preferred treatment protocol
  Arms: Coordinated Care Management Pathway
Behavioral: Nonpharmacological guideline adherent treatment protocol — the pain navigator will select only nonpharmacological guideline adherent treatment options for the patient
  Arms: Coordinated Care Management Pathway
Behavioral: Facilitated referrals to existing VA or non-VA pain management resources — the pain navigator will work with the referring physician to select only existing VA or non-VA pain management resources for the patient.
  Arms: Coordinated Care Management Pathway

SUMMARY:
The purpose and objective of this pragmatic trial is to examine the effectiveness of two different quality improvement care pathways for low back pain (LBP); a sequenced, integrated care pathway (ICP) and 2) a coordinated, care management pathway (CCP). We will test the central hypothesis that the ICP will reduce pain interference with normal activities and improve physical function, as measured by Patient Reported Outcomes Measurement Information System (PROMIS) Short Form scores when compared to the CCP.

ELIGIBILITY:
Clinic eligibility:

* Volunteer and return signed clinic participation agreement
* Availability of clinical personnel willing to deliver the treatment interventions (in either arm).
* Staff and location need to be distinct from other enrolled clinics.
* Clinics can have a variable number of providers, but together meet criteria for range of monthly visits for low back pain.

Participant Survey Eligibility Criteria:

Inclusion Criteria:

1. Age >= 18
2. Seeking care for LBP with or without radiating symptoms from a participating VA primary care clinic
3. Provider determines LBP is appropriate for conservative management
4. Referred to integrated ICP pathway or CCP pathway by participating clinic provider

Exclusion Criteria:

1. Receiving or referred for hospice/ palliative care (defined by encounter codes and CPRS consults)
2. No documented phone number in the electronic health record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1817 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N Hastings, MD, Principal Investigator — Duke University / Durham VA; Steven Z George, PT, PhD, Principal Investigator — Duke University
Locations (1):
- Durham VA, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data sets will be shared a timely manner with privacy and confidentiality protections to facilitate further research, reuse of data, and replication. Publications from this research will be made available to the public through the National Library of Medicine PubMed Central website. To enable broad resource sharing, the study statistician will create de-identified, publication-specific datasets including all variables presented in the publication. The PIs hold responsibility for ensuring that the individuals cannot be re-identified. No data or code that could lead to re-identification of individuals will be released. The analytical datasets and statistical code used will be retained in accordance with VA record retention policy. Study manuals and clinical tools will be shared with the NIH PMC3 Collaboratory and VA health care system facilities. If successful outcomes justify broader dissemination, we will seek to do so by placing relevant materials into the public domain.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data and other resources referenced will be available one year after the date of publication for the primary analyses, which is in alignment with the VA Office of Research and Development.
Access Criteria: We plan on using a de-identified dataset is not subject to HIPAA's minimum necessary standards and would not require a data use agreement. Typically datasets will be provided in SAS transport files using CDISC standards via a website. Requesters will have to enter a valid email, phone number and address to request data. The data provided will be made available under certain requirements and approved on a case by case basis. Requirements include:
  * data will be used for research purposes and not to identify subjects
  * data must be secured using appropriate computer technology
  * data must be destroyed or returned after any analysis are complete
  * authors of any manuscript resulting from this data must acknowledge the source of the data
  * analyses for the purpose of presentations, abstracts, and/or publications must be coordinated through the Publications Committee, to avoid overlap
  * coauthors must be given a chance for review and approval of a draft manuscript prior to submission

REFERENCES:
- [Background] George SZ, Coffman CJ, Allen KD, Lentz TA, Choate A, Goode AP, Simon CB, Grubber JM, King H, Cook CE, Keefe FJ, Ballengee LA, Naylor J, Brothers JL, Stanwyck C, Alkon A, Hastings SN. Improving Veteran Access to Integrated Management of Back Pain (AIM-Back): Protocol for an Embedded Pragmatic Cluster-Randomized Trial. Pain Med. 2020 Dec 12;21(Suppl 2):S62-S72. doi: 10.1093/pm/pnaa348. PMID 33313728
- [Background] Lentz TA, Coffman CJ, Cope T, Stearns Z, Simon CB, Choate A, Gladney M, France C, Hastings SN, George SZ. If You Build It, Will They Come? Patient and Provider Use of a Novel Hybrid Telehealth Care Pathway for Low Back Pain. Phys Ther. 2024 Feb 1;104(2):pzad127. doi: 10.1093/ptj/pzad127. PMID 37756618
- [Background] Ballengee LA, King HA, Simon C, Lentz TA, Allen KD, Stanwyck C, Gladney M, George SZ, Hastings SN. Partner engagement for planning and development of non-pharmacological care pathways in the AIM-Back trial. Clin Trials. 2023 Oct;20(5):463-472. doi: 10.1177/17407745231178789. Epub 2023 Jun 2. PMID 37269070
- [Derived] George SZ, France C, Coffman CJ, Allen KD, Lentz TA, North R, Choate A, Goode AP, Simon CB, Grubber JM, King H, Cook CE, Keefe FJ, Ballengee LA, Naylor J, Brothers JL, Stanwyck C, Linton T, Tumminello C, Hastings SN. Cohort Profile: Baseline Characteristics of Veterans from Improving Veteran Access to Integrated Management of Back Pain (AIM-Back) - an Embedded Pragmatic, Cluster Randomized Trial in the United States. medRxiv [Preprint]. 2024 Nov 26:2024.11.23.24317833. doi: 10.1101/2024.11.23.24317833. PMID 39649618
- See also: Updated Statistical Analysis Plan Preprint — https://www.medrxiv.org/content/10.1101/2023.12.22.23300382v1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A subset of the overall population was recruited to participate in a series of telephone surveys.
Units Other Than Participants: Primary Care Clinics
Period: Overall Study (All Participants)
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Started | 811; 8 Primary Care Clinics | 1006; 9 Primary Care Clinics
Completed | 461; 8 Primary Care Clinics | 537; 9 Primary Care Clinics
Not Completed | 350; 0 Primary Care Clinics | 469; 0 Primary Care Clinics
Not completed — Lost to Follow-up | 350 | 469
Period: Survey Subset
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Started (A subset of the overall population was recruited to participate in a series of telephone surveys.) | 516; 8 Primary Care Clinics | 480; 9 Primary Care Clinics
Completed | 382; 8 Primary Care Clinics | 360; 9 Primary Care Clinics
Not Completed | 134; 0 Primary Care Clinics | 120; 0 Primary Care Clinics
Not completed — Lost to Follow-up | 134 | 120

BASELINE CHARACTERISTICS:
Population: Due to AIM-BACK being a cluster randomized trial design, there is some enrollment variability across clinics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway | Total
Number analyzed (Participants) | 811 | 1006 | 1817
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.4) | 52.7 (15.9) | 53 (15.7)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A subset of the overall participants was recruited to participate in a series of telephone surveys.
  years
    number analyzed (Participants) | 516 | 480 | 996
    (all) | 51.4 (15.1) | 52.0 (15.6) | 51.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 110 | 220
  Male | 701 | 896 | 1597
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A subset of the overall participants was recruited to participate in a series of telephone surveys.
  Participants
    number analyzed (Participants) | 516 | 480 | 996
    Female | 65 | 44 | 109
    Male | 451 | 436 | 887
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 59 | 95
  Not Hispanic or Latino | 766 | 920 | 1686
  Unknown or Not Reported | 9 | 27 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A subset of the overall participants was recruited to participate in a series of telephone surveys.
  Participants
    number analyzed (Participants) | 516 | 480 | 996
    Hispanic or Latino | 37 | 48 | 85
    Not Hispanic or Latino | 476 | 429 | 905
    Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 7 | 11
  Asian | 2 | 10 | 12
  Native Hawaiian or Other Pacific Islander | 4 | 8 | 12
  Black or African American | 301 | 232 | 533
  White | 466 | 703 | 1169
  More than one race | 8 | 16 | 24
  Unknown or Not Reported | 26 | 30 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A subset of the overall participants was recruited to participate in a series of telephone surveys.
  Participants
    number analyzed (Participants) | 516 | 480 | 996
    American Indian or Alaska Native | 5 | 7 | 12
    Asian | 5 | 6 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 166 | 83 | 249
    White | 300 | 326 | 626
    More than one race | 13 | 24 | 37
    Unknown or Not Reported | 27 | 33 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 811 | 1006 | 1817

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference Measure
Description: The PROMIS Short form scores will be collected by the clinical providers within the medical record at baseline and three months to measure pain interference. The pain interference form asks the participant to rate a series of pain related questions on a scale of 1-5 within the past seven days with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. With the revised statistical analysis plan, the patient reported outcomes survey data were used to supplement missing three month follow up data from the medical record, when possible. A higher score indicates greater pain interference.
Time Frame: Baseline, three months post baseline
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 454 | 527
T-score | -2.67 (7.22) | -2.04 (6.73)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Test type: Superiority; p = 0.169, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; Hierarchical linear model fit included random effects for clinic and clinic by time and pre-specified clinic- and patient-level covariates; Mean Difference (Final Values) = -0.59, 97.5% CI 2-sided [-1.55 to 0.37] — Difference is calculated as Integrated Sequenced Care Pathway 3-month change minus Coordinated Care Management Pathway 3-month change

2. Primary Outcome: Change in Physical Function Measure
Description: The PROMIS Short form scores will be collected by the clinical providers within the medical record at baseline and three months to measure physical function. The physical function form asks the participant to rate a series of physical function related questions on a scale of 1-5 within the past seven days with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. With the revised statistical analysis plan, the patient reported outcomes survey data were used to supplement missing three month follow up data from the medical record, when possible. A higher score indicates better physical function.
Time Frame: Baseline, three months post baseline
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 458 | 531
T-score | 1.87 (5.70) | 1.44 (5.14)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Test type: Superiority; p = 0.139, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.59, 97.5% CI 2-sided [-0.33 to 1.52] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Sleep Disturbance
Description: The PROMIS Short form scores will be collected in the medical record by the provider at baseline, and three months post baseline to measure sleep disturbance. The sleep disturbance form asks the participant to rate a series of sleep related questions on a scale of 1-5 with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. With the revised statistical analysis plan, the patient reported outcomes survey data were used to supplement missing three month follow up data from the medical record, when possible. A higher score indicates greater sleep disturbance.
Time Frame: Baseline, three months post baseline
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 456 | 529
T-score | -2.56 (7.35) | -2.06 (8.01)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Test type: Superiority; p = 0.417, Mixed Models Analysis — P-value is not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.69 to 0.72]

4. Secondary Outcome: Change in Patient Reported Outcomes--PROMIS Sleep Disturbance
Description: The PROMIS Short form scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure sleep disturbance. The sleep disturbance form asks the participant to rate a series of sleep related questions on a scale of 1-5 with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. A higher score indicates greater sleep disturbance.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 425 | 414
T-score
  Baseline to 3 months | -1.35 (6.92) | -1.07 (6.60)
  Baseline to 6 months: number analyzed (Participants) | 409 | 384
  Baseline to 6 months | -1.50 (6.65) | -1.66 (6.89)
  Baseline to 12 months: number analyzed (Participants) | 382 | 360
  Baseline to 12 months | -1.25 (7.14) | -1.26 (7.26)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.409, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.37 to 0.57] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.899, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.04 to 0.91] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.946, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.01 to 1.08] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

5. Secondary Outcome: Number of Participants With Opioid Use--Chronic User
Description: Opioid use will be defined at baseline and 12 months post baseline as a binary variable based on whether a chronic opioid user or not at baseline and at twelve months. Opioid use is chronic if participant had at least one prescription with a total day supply of at least 120 days or if there were at least 10 prescription fills in the 12 months prior to the specified timepoint (baseline, 12 months post baseline).
Time Frame: Baseline, twelve months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 811 | 1006
Participants
  Baseline | 28 | 36
  12 months | 22 | 26
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Test type: Superiority; p = 0.992, Regression, Logistic — P-value is not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio, log = -0.004, 95% CI 2-sided [-4.62 to 4.61] — Odds Ratio calculated for Integrated Sequenced Care Pathway relative to Coordinated Care Management Pathway

6. Secondary Outcome: Change in Opioid Use - Morphine Dose
Description: Opioid use--morphine dose will be defined at baseline and 12 months post baseline as a continuous variable measuring morphine equivalents for opioid dose at baseline and twelve months. Change in total milligrams of morphine equivalents (MME) use is reported.
Time Frame: Baseline, twelve months post baseline
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 811 | 1006
MME | -2.62 (36.3) | -2.69 (52.3)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Test type: Superiority; p = 0.262, Mixed Models Analysis — P-value is not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -2.67, 95% CI 2-sided [-7.52 to 2.18] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

7. Secondary Outcome: Change in Patient Reported Outcomes--PROMIS Pain Interference
Description: The PROMIS Short form scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure pain interference. The pain interference form asks the participant to rate a series of pain related questions on a scale of 1-5 within the past seven days with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. A higher score indicates greater pain interference.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 424 | 410
T-score
  Baseline to 3 months | -1.44 (6.19) | -1.10 (6.08)
  Baseline to 6 months: number analyzed (Participants) | 408 | 381
  Baseline to 6 months | -1.64 (6.29) | -1.22 (6.69)
  Baseline to 12 months: number analyzed (Participants) | 381 | 358
  Baseline to 12 months | -1.77 (6.50) | -1.31 (6.65)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.37, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.40, 97.5% CI 2-sided [-1.31 to 0.50] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.24, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 97.5% CI 2-sided [-1.54 to 0.39] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.37, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.45, 97.5% CI 2-sided [-1.43 to 0.54] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

8. Secondary Outcome: Change in Patient Reported Outcomes--PROMIS Physical Function
Description: The PROMIS Short form scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure physical function. The physical function form asks the participant to rate a series of physical function related questions on a scale of 1-5 with 1 representing a better outcome. Ratings are summed across the four questions and converted to a standardized T-score (mean 50, standard deviation 10) according to PROMIS Scoring tables. Observations with 1 missing rating (of 4) were scored using the auto-scoring template in REDCap; observations with more than 1 missing rating were not scored and so were coded as missing. A higher score indicates better physical function.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 424 | 414
T-score
  Baseline to 3 months | -0.20 (4.55) | -0.15 (4.62)
  Baseline to 6 months: number analyzed (Participants) | 408 | 384
  Baseline to 6 months | 0.24 (5.07) | 0.14 (4.83)
  Baseline to 12 months: number analyzed (Participants) | 382 | 359
  Baseline to 12 months | -0.09 (5.02) | 0.08 (5.17)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.727, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.11, 97.5% CI 2-sided [-0.51 to 0.72] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.478, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.24, 97.5% CI 2-sided [-0.43 to 0.91] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.894, Mixed Models Analysis — Threshold for significance is 0.025 due to dual primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 97.5% CI 2-sided [-0.75 to 0.66] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

9. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Catastrophizing
Description: Catastrophizing questions from the NIH recommended minimum data set will be collected by the interviewers at baseline, three, six, and twelve months post baseline and will evaluate catastrophizing with two agree (1) / disagree (0) questions. Responses marked as DK/Ref/Missing are coded as missing. Responses are then summed across the two questions; possible outcome values are 0, 1, 2. A higher score indicates greater catastrophizing.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 352 | 303
score on a scale
  Baseline to 3 months: number analyzed (Participants) | 338 | 303
  Baseline to 3 months | 0.08 (0.66) | 0.08 (0.71)
  Baseline to 6 months: number analyzed (Participants) | 352 | 275
  Baseline to 6 months | 0.11 (0.62) | 0.07 (0.76)
  Baseline to 12 months: number analyzed (Participants) | 309 | 267
  Baseline to 12 months | 0.05 (0.72) | 0.09 (0.77)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.222, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.15 to 0.04] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.988, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.10 to 0.09] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.269, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.16 to 0.05] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

10. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Alcohol Use Disorders Identification Test Concise (AUDIT-C)
Description: The AUDIT-C form scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure alcohol use. The AUDIT-C form asks the participant to rate three alcohol use questions on a scale of 0-4 with zero representing a better outcome. The total score is the sum of the non-missing responses to the three questions, with range of possible values 0-12.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 425 | 414
score on a scale
  Baseline to 3 months | -0.17 (1.11) | -0.14 (1.36)
  Baseline to 6 months: number analyzed (Participants) | 409 | 384
  Baseline to 6 months | -0.17 (1.35) | -0.19 (1.37)
  Baseline to 12 months: number analyzed (Participants) | 382 | 360
  Baseline to 12 months | -0.25 (1.46) | -0.18 (1.49)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.477, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.22 to 0.10] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.877, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.19 to 0.17] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.360, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.29 to 0.11] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

11. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Pain Intensity, Enjoyment of Life, General Activity (PEG) Screening Tool
Description: The PEG screening tool scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure pain intensity. The PEG form asks the participant to rate a series of pain intensity related questions on a scale of 0-10 with 0 representing a better outcome. The total score is the sum of responses to the three questions and is missing if any of the three questions is missing. The range of possible values is 0-30.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 422 | 411
score on a scale
  Baseline to 3 months | -0.35 (1.89) | -0.42 (1.94)
  Baseline to 6 months: number analyzed (Participants) | 405 | 382
  Baseline to 6 months | -0.44 (1.94) | -0.42 (2.05)
  Baseline to 12 months: number analyzed (Participants) | 378 | 357
  Baseline to 12 months | -0.38 (2.09) | -0.38 (2.15)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.858, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.23 to 0.28] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.688, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.32 to 0.21] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.833, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.32 to 0.26] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

12. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Pain Self Efficacy Questionnaire (PSEQ-2)
Description: Pain Self-Efficacy Questionnaire from the PSEQ-2 form will be collected by the interviewers at baseline, three, six, and twelve months post baseline and will evaluate self-efficacy on a scale of 0-6 with zero representing a worse outcome. The total score is the sum of responses to the two questions and is missing if either of the two questions is missing. The range of possible values is 0-12.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 409 | 391
score on a scale
  Baseline to 3 months | -0.13 (2.82) | -0.38 (3.02)
  Baseline to 6 months: number analyzed (Participants) | 395 | 365
  Baseline to 6 months | -0.08 (2.73) | -0.46 (2.98)
  Baseline to 12 months: number analyzed (Participants) | 369 | 343
  Baseline to 12 months | -0.22 (2.88) | -0.39 (2.90)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.259, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.18 to 0.64] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.068, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.03 to 0.81] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.514, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.29 to 0.57] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

13. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Depressed Mood
Description: The Patient Health Questionnaire-2 (PHQ2) form scores will be collected by the interviewers at baseline, three, six, and twelve months post baseline to measure depressed mood. The PHQ2 form asks the participant to answer two questions about potential depressed mood within the past week with ratings between 0 and 3. The total score is the sum of responses to the two questions and is missing if either of the two questions is missing. The range of possible values is 0-6. A higher score indicates greater depressed mood.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 416 | 404
score on a scale
  Baseline to 3 months | 0.02 (1.44) | 0.04 (1.60)
  Baseline to 6 months: number analyzed (Participants) | 403 | 375
  Baseline to 6 months | 0.09 (1.58) | 0.02 (1.58)
  Baseline to 12 months: number analyzed (Participants) | 376 | 355
  Baseline to 12 months | -0.01 (1.57) | 0.02 (1.60)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.895, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.22 to 0.20] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.438, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.13 to 0.30] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.890, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.24 to 0.21] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

14. Other Pre Specified Outcome: Change in Patient Reported Outcomes--Quality of Life
Description: The EuroQoL five-item quality of life questionnaire, EQ-5D-5L, will be administered by interviewers at baseline, three, six, and twelve months post baseline to measure quality of life. The EQ-5D-5L asks the participant five questions related to quality of life on a scale of 1-5. If all questions are answered, the responses are concatenated to form a 5-digit state in the order mobility, self care, usual activities, pain discomfort, anxiety/depression. This 5-digit state is then converted to an index between 0 and 1. A higher score indicates greater quality of life.
Time Frame: Baseline, three, six, and twelve months
Population: Participants with data collected collected at both timepoints needed to calculate a change.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
Number analyzed (Participants) | 415 | 405
score on a scale
  Baseline to 3 months | -0.04 (0.26) | -0.03 (0.25)
  Baseline to 6 months: number analyzed (Participants) | 404 | 377
  Baseline to 6 months | 0.04 (0.26) | -0.04 (0.25)
  Baseline to 12 months: number analyzed (Participants) | 379 | 354
  Baseline to 12 months | -0.04 (0.26) | -0.02 (0.26)
Statistical Analysis 1: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 3 months; Test type: Superiority; p = 0.508, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.01, 95% CI 2-sided [-0.04 to 0.02] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 2: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 6 months; Test type: Superiority; p = 0.992, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.03 to 0.03] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change
Statistical Analysis 3: Comparison: Integrated Care Pathway vs Coordinated Care Management Pathway; Baseline to 12 months; Test type: Superiority; p = 0.389, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. Threshold for significance is 0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.02] — Difference is calculated as Integrated Sequenced Care Pathway change minus Coordinated Care Management Pathway change

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Adverse Events were collected on survey participants only. A non-systematic method was implemented. Adverse events were collected via unsolicited participant self-report during follow-up study surveys. Study staff attempted to verify reported adverse events via medical record review. All hospitalizations were considered serious and Emergency Department visits were considered important medical events. All events were assessed for study relatedness. All events were reviewed by the Durham VA IRB.
Arm/Group | Integrated Care Pathway | Coordinated Care Management Pathway
All-Cause Mortality (participants affected / at risk) | 1/516 | 2/480
Serious Adverse Events (participants affected / at risk) | 18/516 | 30/480
Other Adverse Events (participants affected / at risk) | 12/516 | 20/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Care Pathway (N=516) | Coordinated Care Management Pathway (N=480)
Hospitalization (General disorders) | 18 (18) | 30 (30)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Care Pathway (N=516) | Coordinated Care Management Pathway (N=480)
Important Medical Events (General disorders) | 12 (12) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT04411420/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04411420/ICF_001.pdf